CLINICAL TRIAL: NCT07276971
Title: The Effect of the Safe Early Mobilization Protocol Developed for Patients Underwent Coronary Artery Bypass Graft Surgery on Patient Outcomes
Brief Title: The Safe Early Mobilization on CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hulya BULUT (Other)
Collaborators: Lokman Hekim University (Other Government); Ankara Guven Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Hulya BULUT, Prof. Dr., Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 36970
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Bypass Graft; Nursing
Keywords: Coronary artery bypass graft; Cardiovascular nursing; Early mobilization protocol; Patient outcomes
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEMP (Experimental): A safe early mobilization protocol developed by the researchers was applied.
  Interventions: Other: The safe early mobilization protocol
- Control group (Active Comparator): The routine protocol used in the hospital was applied.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: The safe early mobilization protocol — This protocol was developed to guide the early postoperative mobilization of patients undergoing coronary artery bypass graft surgery, covering the period from the day of surgery to the fourth postoperative day. Prior to mobilization, patients are evaluated using a checklist ensuring physical and environmental safety. On the day of surgery, following extubation by the responsible physician, six stages are applied: bed head elevation, deep breathing exercises, incentive spirometry, passive range of motion (ROM) exercises, sitting upright (90°), and sitting on the edge of the bed. On postoperative days 1-3, standing at the bedside, ambulation, and sitting on a chair are added. Target walking distances are 100-150 m on day 1, 200-250 m on day 2, and 300-350 m on day 3. Distances are measured by the researcher using a meter. The protocol concludes on the 4th postoperative day when the patient can ambulate independently.
  Arms: SEMP
Other: Control Group — Patients in the control group were informed about the current mobilization practices applied in the clinic before surgery. The morning after the surgery (the first day after the surgery), the patient is first seated in the bed, and in the second stage, he is made to sit on the edge of the bed with his feet touching the floor and is observed. In the third stage, the patient stands in an upright position and if there is no dizziness or blackout, the patient is seated on a chair next to the bed. The duration of sitting in the chair is determined depending on the general condition of the patient (pain, dizziness, blackout, nausea). On the 2nd and 3rd postoperative day, patients were contacted by nurses and care support staff while they had a chest tube; Then, the patient is mobilized only with his/her relative. There is no standard practice regarding how long patients should be mobilized during the day.
  Arms: Control group

SUMMARY:
Aim: This study aimed to evaluate the effect of a Safe Early Mobilization Protocol (SEMP) developed for patients undergoing coronary artery bypass graft (CABG) surgery on patient outcomes.

Design: A single-center, parallel-group, randomized controlled trial. Methods: The study was conducted with 60 patients in 2023. The intervention group received a Safe Early Mobilization Protocol including bedside elevation, deep breathing and coughing exercises, sitting upright in bed, sitting on the edge of the bed, standing, ambulation, and sitting in a bedside chair from the day of surgery until the fourth postoperative day. The control group received routine mobilization care. Respiratory parameters, orthostatic hypotension (OH), orthostatic intolerance (OI), mobilization distance, anxiety level, and hospital stay were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Hemodynamic stability, defined as:

Resting heart rate <110/min

Mean arterial pressure between 60-110 mmHg

Oxygen saturation (SpO₂) >88%

Receiving dopamine infusion ≤5 mcg/kg/min at the time of enrollment

No auditory, speech, or visual impairments

No neurological contraindications (e.g., cerebrovascular accident [CVA], ataxia, multiple sclerosis [MS])

No orthopedic contraindications that prevent mobilization (e.g., fractures or sequelae)

Provided informed consent to participate in the study

Age ≥18 years

Able to speak Turkish

Literate patients

Exclusion Criteria:

Requirement for intra-aortic balloon pump (IABP) support

Postoperative cerebrovascular events

High-dose inotropic drug infusion in the early postoperative period:

Dopamine ≥10 mcg/kg/min

Norepinephrine ≥0.5 mcg/kg/min

Concurrent dopamine and norepinephrine infusion

Severe arrhythmias preventing mobilization, including:

Sinus tachycardia ≥120/min

Rapid atrial fibrillation

Ventricular tachycardia

Ventricular fibrillation

Advanced chronic obstructive pulmonary disease (COPD) or bronchiectasis

Diagnosed anxiety disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Orthostatic Hypotension | Daily postoperative measurements for up to 3 days.
  Orthostatic hypotension defined as a ≥20 mmHg decrease in systolic BP and/or ≥10 mmHg decrease in diastolic BP.
Number of Participants With Orthostatic Intolerance | Daily postoperative assessments for up to 3 days.
  Orthostatic intolerance defined as the presence of dizziness, nausea, weakness, blurred vision, or syncope.considered as OI.
Oxygen Saturation Level (%) | Daily postoperative measurements for up to 3 days.
  Peripheral oxygen saturation (SpO₂) measured using pulse oximetry.
State Anxiety Scale Score | Postoperative day 1 and postoperative day 4.
  The State Anxiety Inventory (STAI-S) will be used (score range: 20-80; higher scores indicate worse anxiety).
Six-Minute Walk Test Distance (Meters) | Postoperative day 4.
  Distance walked during the Six-Minute Walk Test (0-∞ meters; higher distance indicates better functional capacity).

SECONDARY OUTCOMES:
Length of Hospital Stay (Days) | From postoperative day 0 until hospital discharge (up to 30 days).
  Total duration of postoperative hospitalization, including ICU and ward stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Guven Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared when the study is published.